CLINICAL TRIAL: NCT04211623
Title: Comparison of Constrained Induced Movement Therapy and Bimanual Intensive Movement Therapy on Functional Outcome of Hemiplegic Cerebral Palsy
Brief Title: CIMT and BIMT Affect Functional Outcome in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIUHumaile
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Cerebral Palsy, Congenital
Keywords: Cerebral Palsy; Neurorehabilitation; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint induced movement therapy group (Active Comparator): Constrained on more affected side for three hours.
  Interventions: Other: Constraint induced movement therapy
- Bimanual activities group; BIM training (Active Comparator): Set of bimanual activities performed.
  Interventions: Other: Bimanual activities

INTERVENTIONS:
Other: Constraint induced movement therapy — Constrained on more affected side for three hours. To minimize the learned non use in hemiplegic CIMT is applied and criteria of applying CIMT is;
  * 10 degrees active wrist extension on the affected hand,
  * 10 degrees active thumb abduction,
  * 10 º active extension of any two digits on the side or hand which is limited due to damage.
  In order to gain the maximum good results from CIMT technique following points should also be considered attentively. Affected arm should move to 45 degrees shoulder flexion and abduction, and 90 degrees of elbow flexion and extension.
  Constrained with cotton sling. 3 to 5 upper limb functional activities like
  * using fork or a spoon,
  * combing hair
  * brushing teeth
  * writing
  * dressing all activities are performed for 10 t0 15 minutes in period of three hours on alternate days in a week
  Arms: Constraint induced movement therapy group
Other: Bimanual activities — Bimanual activities of both hands are performed like
  Set of bimanual activities is used to assess the bimanual hand function. Five bimanual activities are performed such as
  * carrying a tray,
  * cutting a fruit with a knife,
  * holding and cutting the paper with scissor,
  * buttoning and
  * Carrying heavy objects with both hands.
  Every activity was performed for 10 t0 15 minutes on alternate days for a period of 6 weeks session.
  Arms: Bimanual activities group; BIM training

SUMMARY:
The aim of this randomized controlled trial is to determine the effects of constraint induced movement therapy CIMT and BIM bimanual activities on functional outcome in hemiplegic CP. Two randomized groups of patients with CP are treated with constrained arm for three hours on affected side and bimanual activities on BIM group respectively. Both, male and female patients meeting the inclusion criteria will be included. Patients having concurrent malignancy, infection, trauma or any bony deformity will be excluded.

DETAILED DESCRIPTION:
It is a Randomized control trial. Cerebral palsy children of age groups of 5 yrs to 12 years were included in the study with total sample size of thirty eight (38) with confidence interval of 95%. Simple random sampling was done by lottery method and data was collected from ALFARABI special school of education Islamabad. Two groups were formed and named as group A; CIMT with nineteen participants and group B, BIM bimanual training with nineteen participants respectively. The RCT compared the functional outcome of 3 hours constraining for 3 times a week for 6 weeks duration for CIMT group and five bimanual activities performed for three hours a day for bimanual group B and were assessed on the pretest and post test score evaluation of QUEST and JTHF test. All the participants were hemiplegic cp from both gender, fall on MAC system level II. Treatment for three hours was done on alternate days for 3 days a week. Five bimanual activites of holding a tray, cutting a fruit with knife, buttoning, cutting paper with scissor, and carry heavy objects with both hands are applied. Whereas the activities performed in CIMT are brushing teeth, holding spoon, fork combing hair and writing. Forty five children were screened before the evaluation and as a result 38 were enrolled in both groups having 19 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age group of 5-12 years. Patients with hemiplegic cerebral palsy of both genders. Patients who have active wrist extension, active PIP -MCP joint extension and active thumb extension.

Patients who have mild spasticity on spasticity rating scale of QUEST test Patients who fall on level II on MAC System are included Patients who has cognitive dysfunction ( screening by WISC Wechsler Intelligence test for children) all have score above 80.

Exclusion Criteria:

* Patients who can develop any sort of behavior problems Patients who does not co-operate with therapist in CIMT procedure Any structural deformity. Any surgical intervention that requires patient to be immobile.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Quality of upper extremity skills test | 6 weeks
  Quality of upper extremity skills test or QOL quality of life. This scoring includes dissociated movements, grasps, weight bearing and protected extension. This scoring helps the therapist to determine which functional limitations needs to be addressed for better flexion extension abduction and other related movements to improve quality of life . It includes 36 items to be tested and thirty to forty minutes to apply and assess the test.
JEBSEN Hand Function Test | 6 weeks
  The JEBSEN Hand Function Test was designed to provide a comprehensive, objective test of hand function for actions of daily living. It has 7 items and takes approximately 15-45 minutes to administer. 7 items include: writing, turning over 3-by-5 inch cards, picking up small common objects, stacking checkers, simulated feeding, picking up large light objects and picking up large heavy objects. The results are calculated by timing the time taken to complete each task. The tests are always presented in the same order and are performed with the non-dominant hand first

SECONDARY OUTCOMES:
Manual ability classification | 6 weeks
  The Manual Ability Classification System (MACS) describes how children with (CP) use their hands to carry objects in daily routine. MAC describes 5 levels. These levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life. The MACS also describe differences between adjacent levels to make it easier to determine which level best corresponds with the child's capability to handle objects. The objects are relevant and age-appropriate for the children, used when they perform tasks such as eating, dressing, playing, drawing or writing. Etc.

CONTACTS AND LOCATIONS:
Overall Officials: Mir Arif Hussain, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charles J, Gordon AM. Development of hand-arm bimanual intensive training (HABIT) for improving bimanual coordination in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2006 Nov;48(11):931-6. doi: 10.1017/S0012162206002039. PMID 17044964
- [Background] Charles J, Gordon AM. A critical review of constraint-induced movement therapy and forced use in children with hemiplegia. Neural Plast. 2005;12(2-3):245-61; discussion 263-72. doi: 10.1155/NP.2005.245. PMID 16097492
- [Background] Sakzewski L, Ziviani J, Boyd R. Systematic review and meta-analysis of therapeutic management of upper-limb dysfunction in children with congenital hemiplegia. Pediatrics. 2009 Jun;123(6):e1111-22. doi: 10.1542/peds.2008-3335. Epub 2009 May 18. PMID 19451190
- [Background] Gordon AM, Schneider JA, Chinnan A, Charles JR. Efficacy of a hand-arm bimanual intensive therapy (HABIT) in children with hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2007 Nov;49(11):830-8. doi: 10.1111/j.1469-8749.2007.00830.x. PMID 17979861
- [Background] Dickerson AE, Brown LE. Pediatric constraint-induced movement therapy in a young child with minimal active arm movement. Am J Occup Ther. 2007 Sep-Oct;61(5):563-73. doi: 10.5014/ajot.61.5.563. PMID 17944294
- [Background] Geerdink Y, Lindeboom R, de Wolf S, Steenbergen B, Geurts AC, Aarts P. Assessment of upper limb capacity in children with unilateral cerebral palsy: construct validity of a Rasch-reduced Modified House Classification. Dev Med Child Neurol. 2014 Jun;56(6):580-6. doi: 10.1111/dmcn.12395. Epub 2014 Feb 11. PMID 24517893
- [Background] Dong VA, Tung IH, Siu HW, Fong KN. Studies comparing the efficacy of constraint-induced movement therapy and bimanual training in children with unilateral cerebral palsy: a systematic review. Dev Neurorehabil. 2013;16(2):133-43. doi: 10.3109/17518423.2012.702136. Epub 2012 Sep 4. PMID 22946588
- [Background] Obladen M. Lame from birth: early concepts of cerebral palsy. J Child Neurol. 2011 Feb;26(2):248-56. doi: 10.1177/0883073810383173. Epub 2010 Dec 30. PMID 21193777
- [Background] Rosenbaum P, Stewart D. The World Health Organization International Classification of Functioning, Disability, and Health: a model to guide clinical thinking, practice and research in the field of cerebral palsy. Semin Pediatr Neurol. 2004 Mar;11(1):5-10. doi: 10.1016/j.spen.2004.01.002. PMID 15132248
- [Background] Utley A, Steenbergen B, Sugden DA. The influence of object size on discrete bimanual co-ordination in children with hemiplegic cerebral palsy. Disabil Rehabil. 2004 May 20;26(10):603-13. doi: 10.1080/09638280410001696674. PMID 15204514
- [Background] de Brito Brandao M, Mancini MC, Vaz DV, Pereira de Melo AP, Fonseca ST. Adapted version of constraint-induced movement therapy promotes functioning in children with cerebral palsy: a randomized controlled trial. Clin Rehabil. 2010 Jul;24(7):639-47. doi: 10.1177/0269215510367974. Epub 2010 Jun 8. PMID 20530645
- [Background] Wittenberg GF, Schaechter JD. The neural basis of constraint-induced movement therapy. Curr Opin Neurol. 2009 Dec;22(6):582-8. doi: 10.1097/WCO.0b013e3283320229. PMID 19741529